CLINICAL TRIAL: NCT01570413
Title: Utility of Pelvic Examination in the Evaluation of Threatened Abortion
Brief Title: Pelvic Examination in Pregnancy
Acronym: PEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Principal Investigator, Judith Linden, BMC Faculty, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: H-31421
Record Dates: First submitted 2012-02-27; First posted 2012-04-04 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Early Pregnancy Bleeding; Abdominal Pain
MeSH Terms: conditions — Abdominal Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pelvic Exam (Active Comparator): Subjects receive pelvic exam
  Interventions: Procedure: Pelvic Examination
- No Pelvic Exam (Experimental): Subjects do not receive pelvic exam
  Interventions: Procedure: No Pelvic Exam

INTERVENTIONS:
Procedure: No Pelvic Exam — Will not receive pelvic examination.
  Arms: No Pelvic Exam
Procedure: Pelvic Examination — Pelvic examination will be performed.
  Arms: Pelvic Exam

SUMMARY:
This study is designed to determine whether the pelvic examination (including bimanual and speculum examination) is necessary in patients with first trimester vaginal bleeding/ lower abdominal pain when an intra-uterine pregnancy (IUP) is seen on ultrasound. Patients with the chief complaint of vaginal bleeding or lower abdominal pain less than 16 weeks and positive HCG will be considered for this non-inferiority-designed clinical trial. All patients who present to the BMC Emergency Department (ED) Mon - Fri from 8am to 11pm and have had serum or urine HCG testing and a formal ultrasound by a credentialed emergency physician or radiology technician as part of standard of care will be screened for further eligibility. Those patients with intra-uterine pregnancies < 16 weeks gestation seen on ultrasound and meet inclusion criteria will then be asked to provide informed consent to participate in the study. Randomization will occur after consent has been obtained. Half of the patients will be randomized to receive pelvic examinations and the other half will not. Further care will be determined by the treating attending physician. The primary outcome will be a composite morbidity endpoint at 30 days, including return visits to the ED, emergency surgery, need for transfusion, infection, or other missed source of bleeding/ pain. Secondary outcomes of interest include ED throughput time, and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

1. Chief complaint of vaginal bleeding or lower abdominal pain
2. Intra-uterine pregnancy seen on ultrasound
3. Date < 16 weeks by estimated LMP or ultrasound
4. Age >21
5. Ability to provide written informed consent
6. English speaking

Exclusion Criteria:

1. Already enrolled in study
2. Morbid Obesity (BMI > 40)
3. Pelvic exam performed prior to ultrasound results
4. Prisoner
5. Follow up cannot be assured
6. Admitted to hospital
7. Large amount of vaginal bleeding (>10 pads in 24 hours or equivalent)
8. Unstable vital signs (SBP<90 or HR>110)
9. Known cervical carcinoma in the past 1 year
10. Clinical suspicion for alternative syndrome that requires pelvic exam (such as severe pain consistent with ovarian torsion)
11. Report or suspicion of penetrating vaginal trauma
12. Suspicion of Active Labor
13. Reported Sexual Assault
14. Current pregnancy by IVF
15. IUD in place
16. Suspicion of heterotopic pregnancy on ultrasound

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2012-02; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Composite Morbidity Endpoint | 30 Days
  Adverse events include, but are not limited to, return visits to the Emergency Department, need for hospital admission, emergency procedure, transfusion, infection, or identification of other source of symptoms.

SECONDARY OUTCOMES:
Patient Satisfaction | 24 Hours
Throughput Time | 24 Hours

CONTACTS AND LOCATIONS:
Overall Officials: Judith Linden, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Brown J, Fleming R, Aristzabel J, Gishta R. Does pelvic exam in the emergency department add useful information? West J Emerg Med. 2011 May;12(2):208-12. PMID 21691528
- [Background] Brown T, Herbert ME. Medical myth: Bimanual pelvic examination is a reliable decision aid in the investigation of acute abdominal pain or vaginal bleeding. CJEM. 2003 Mar;5(2):120-2. doi: 10.1017/s1481803500008289. PMID 17475104
- [Background] Hoey R, Allan K. Does speculum examination have a role in assessing bleeding in early pregnancy? Emerg Med J. 2004 Jul;21(4):461-3. doi: 10.1136/emj.2003.012443. PMID 15208231
- [Background] Isoardi K. Review article: the use of pelvic examination within the emergency department in the assessment of early pregnancy bleeding. Emerg Med Australas. 2009 Dec;21(6):440-8. doi: 10.1111/j.1742-6723.2009.01227.x. PMID 20002713
- [Background] Seymour A, Abebe H, Pavlik D, Sacchetti A. Pelvic examination is unnecessary in pregnant patients with a normal bedside ultrasound. Am J Emerg Med. 2010 Feb;28(2):213-6. doi: 10.1016/j.ajem.2008.10.018. PMID 20159393